CLINICAL TRIAL: NCT00005337
Title: Hostility and Coronary Risk--Role of Weak Vagal Function
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4196; R01HL044998 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia

SUMMARY:
To determine whether deficient vagal antagonism of sympathetic nervous system (SNS) actions on the heart contributed to increased coronary heart disease risk in hostile persons.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Sophisticated electrophysiologic monitoring approaches were used to: 1) show greater sensitivity in nonhostile young men to T-wave attenuation effects of isoproterenol infusion following vagal blockade; 2) show that vagal enhancement reduced and shortened the T-wave attenuation effects of isoproterenol infusion more in hostile young men; 3) evaluate these effects of vagal blockage and enhancement in middle-aged men and in young and middle-aged women; and 4) relate the T-wave effects in these studies to other measures of vagal tone and other biobehavioral mechanisms of coronary-prone behavior.

Four studies were conducted in normal young and middle-aged men and women selected as high and low on hostility, evaluating vagal tone measures and effects of isoproterenol infusion on EKG T-wave and ST response after pretreatment with saline, neostigmine, and atropine. Demonstration that hostility was associated with deficient vagal anatagonism of SNS effects on the heart, especially in middle-aged as compared to younger persons, suggested that diminished vagal tone was one pathway whereby high hostility contributed to increased CHD risk. Clinical studies were then conducted to determine whether weaker vagal tone predicted increased myocardial ischemia and/or poorer outcomes in coronary heart disease patients.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-04; Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Redford Williams — Duke University

REFERENCES:
- [Background] Williams RB. Lower socioeconomic status and increased mortality: early childhood roots and the potential for successful interventions. JAMA. 1998 Jun 3;279(21):1745-6. doi: 10.1001/jama.279.21.1745. No abstract available. PMID 9624030
- [Background] Williams RB. The mind, the body, health, and disease. What do we know, what should we do? N C Med J. 1998 May-Jun;59(3):172-4. No abstract available. PMID 9610159
- [Background] Barefoot JC, Helms MJ, Mark DB, Blumenthal JA, Califf RM, Haney TL, O'Connor CM, Siegler IC, Williams RB. Depression and long-term mortality risk in patients with coronary artery disease. Am J Cardiol. 1996 Sep 15;78(6):613-7. doi: 10.1016/s0002-9149(96)00380-3. PMID 8831391
- [Background] Fukudo S, Lane JD, Anderson NB, Kuhn CM, Schanberg SM, McCown N, Muranaka M, Suzuki J, Williams RB Jr. Accentuated vagal antagonism of beta-adrenergic effects on ventricular repolarization. Evidence of weaker antagonism in hostile type A men. Circulation. 1992 Jun;85(6):2045-53. doi: 10.1161/01.cir.85.6.2045. PMID 1317272
- [Background] Williams RB. Hostility and heart disease: Williams et al. (1980). Adv Mind Body Med. 2001 Winter;17(1):52-5. No abstract available. PMID 11270067